CLINICAL TRIAL: NCT00063609
Title: The Effect of Zoledronic Acid Compared to Placebo on Bone Mineral Density in Patients Undergoing Androgen Deprivation Therapy
Brief Title: The Effect of Zoledronic Acid on Bone Loss in Prostate Cancer Patients Undergoing Androgen Deprivation Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CZOL446GUS45; ZENITH
Record Dates: First submitted 2003-07-01; First posted 2003-07-03 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Bone Loss; Osteoporosis; Bone Mineral Density; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Bone Diseases, Metabolic; Osteoporosis | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
The purpose of this study is to compare the effect of an investigational drug used intravenously and placebo administered every three months for one year, on bone loss associated with initial androgen deprivation) in men with prostate cancer without metastasis. In order to participate in this trial male patients must be 18 years of age or older and have been diagnosed with prostate cancer without metastasis and within one year of starting their androgen deprivation therapy at the day of randomization onto this trial. In addition, patients who have undergone a recent orchiectomy (or"ke-ek'te-me) (removal of one or two testes) are eligible to participate.

Patients who received any prior bisphosphonate therapy or prior treatment with systemic corticosteroids within in the past 12 months are not eligible to participate. Also patients who are receiving treatment for osteoporosis are not eligible to participate.

Inclusion into this clinical trial with this investigational drug is based on the protocol entry criteria and evaluation from a participating trial investigator.

ELIGIBILITY:
* Histologically confirmed diagnosis of carcinoma of the prostate
* No distant metastases (stage TNMO) (ie. prostate cancer without metastases)
* Patients within one year at the day of randomization from initiation of androgen deprivation therapy with a LHRH agonist (with or without an antiandrogen) and with the intended duration of androgen deprivation therapy of at least 12 months. Patients may also enter if they have received an orchiectomy (or"ke-ek'te-me) within two weeks of visit 1
* Patients who received any prior bisphosphonate therapy in the past 12 months will be excluded
* Patients who are currently receiving diethylstilbesterol (DES) or PC-SPES (treatment for osteoporosis) will be excluded
* Patients who have received prior treatment with systemic corticosteroids within the past 12 months will be excluded (short term corticosteroid therapy, e.g. to prevent/treat chemotherapy-induced nausea/vomiting or for acute illness like asthma exacerbation, is acceptable)
* Other eligibility criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-04; Study Completion 2005-04

PRIMARY OUTCOMES:
Percent change in bone mineral density of the lumbar spine (L2-L4) at one year.

SECONDARY OUTCOMES:
Percent changes in bone mineral density of the total hip
biochemical markers of bone turnover at one year

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Millennium Therapeutics & Research, Birmingham, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Donald Gleason, MD, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Advanced Urology Med. Center, Anaheim, California
  - Atlantic Urological Medical Group, Long Beach, California
  - San Diego Uro. Research, San Diego, California
  - Western Clinical Research, Torrance, California
  - Connecticut Surgical Group, Hartford, Connecticut
  - Grove Hill Urology, New Britain, Connecticut
  - Atlantic Urological Associates, Daytona Beach, Florida
  - University of Miami School of Medicine, Dept. of Urology, Miami, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Urosearch, Ocala, Florida
  - Southeastern Urological Center, PA, Tallahassee, Florida
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - The Iowa Clinic, PC, Iowa Urology Research, Des Moines, Iowa
  - Summitt Clinical Research, Owings Mills, Maryland
  - Millennium Medical Center, Southfield, Michigan
  - Quality Clinical Research LLC, Springfield, Nebraska
  - Associated Urologic Specialist, PA, Marlton, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Associates In Urology, LLC, West Orange, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Urological Surgeons of L.I., Garden City, New York
  - Staten Island Urological Research, PC, Staten Island, New York
  - The Urology Group, Cincinnati, Ohio
  - Urological Associates, Inc., Columbus, Ohio
  - Mount Vernon Urological Associates, Mount Vernon, Ohio
  - Oregon Urology Specialists, Eugene, Oregon
  - The Urology Clinic, Portland, Oregon
  - Urologic Associates of Allentown, Allentown, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Triangle Urological Group, Pittsburgh, Pennsylvania
  - Urologic Surgeons of New England, P.C., Providence, Rhode Island
  - University Urological Research Institute, Providence, Rhode Island
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Integrity Clinical Research, LLC, Germantown, Tennessee
  - Urology San Antonio Research, San Antonio, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Seattle Urological Associates, Seattle, Washington
  - Rockwood Clinic, Spokane, Washington